CLINICAL TRIAL: NCT05740488
Title: Efficacy and Safety of Apalutamide in Combination With 89Sr as Neoadjuvant Therapy in Prostate Cancer With ≤10 Bone Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Principal Investigator, Binshen Chen, associate chief physician, Zhujiang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-241-02
Record Dates: First submitted 2023-02-08; First posted 2023-02-23 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer With ≤10 Bone Metastases
MeSH Terms: interventions — apalutamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apalutamide combined with 89Sr and ADT (Experimental): Neoadjuvant therapy with apalutamide in combination with 89Sr and ADT
  Interventions: Drug: Apalutamide; Drug: 89Sr; Drug: Luteinizing Hormone-Releasing Hormone Analog

INTERVENTIONS:
Drug: Apalutamide — 240mg, po, qd
Drug: 89Sr — 100~150MBq(based on weight), iv, q90d
Drug: Luteinizing Hormone-Releasing Hormone Analog — sc, 3.6mg, q30d or 10.8mg, q90d

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of apalutamide in combination with 89Sr as neoadjuvant therapy in prostate cancer with ≤10 bone metastases. The primary endpoint is PFS and the second endpoints are pCR, rPFS, PSA response, pain score, number and extent of bone metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Prostate cancer confirmed by pathological findings;
2. Bone metastasis confirmed by bone scan, the number of bone metastases ≤10
3. Agreement to undergo laparoscopic radical prostatectomy + pelvic lymphadenectomy;
4. ECOG score of 0 - 1
5. Agreement to undergo preoperative and postoperative endocrine therapy and 89Sr radionuclide therapy;
6. Voluntary signing of an ICF for the clinical trial

Exclusion Criteria:

1. Any other tumor disease requiring treatment;
2. Any organ metastasis confirmed by imaging, such as liver and brain metastases, or the possibility of paralysis due to spinal cord metastasis;
3. A history of epilepsy or any condition that may lead to seizures;
4. Severe liver or kidney dysfunction, severe cardiovascular or cerebrovascular diseases, and systemic immune system diseases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 2 years after radical prostatectomy
  progression-free survival

SECONDARY OUTCOMES:
pCR | Up to 1 year
  pathological complete response
rPFS | Up to 3 years
  radiographic progression-free survival
PSA response rate | Up to 3 years
  more than 50% decrease from baseline
pain score | Measured at baseline and follow up visits throughout the study, an average of 3 years
  Measurement of pain assessed by a Visual Analogue Scale (VAS). The analogous visual scale used for this study measures from 0 to 10 the intensity of pain with a series of "faces" that show the intensity in the pain experimentation with categories such as "No pain" in number 0, mild in number 1-3, moderate in number 4-6, intense in number 7-9 and worst in number 10.
number and extent of bone metastases | Up to 3 years
  Bone Scan

CONTACTS AND LOCATIONS:
Overall Officials: Chen Binshen, Study Chair — Southern Medical University, China
Locations (1):
- zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong, China